CLINICAL TRIAL: NCT01074788
Title: Mind Body Therapy During Geriatric Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yaffa Lerman and Shahar Lev-Ari, Tasmc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: tasmc-09-yl-0488; tasmc0488-09 (Other: tasmc)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Patients Who Are in Need of Short or Long Term Rehabilitation Due to Neurological Event (Mainly Stroke) or Post Orthopedic Surgery
Keywords: rehabilitation; mind body therapy; integrative medicine
MeSH Terms: interventions — Mind-Body Therapies

ARMS (1):
- mind body intervention group (Experimental)
  Interventions: Behavioral: mind body therapy

INTERVENTIONS:
Behavioral: mind body therapy — mind-body therapy includes guided imagery, relaxation techniques, mediation and touch therapy.

SUMMARY:
The main goal of geriatric rehabilitation following an acute illness is rapid restoration of normal activity. The key elements are pain control, restoration of bowel functions, good sleep quality, appetite and general well-being, as well as return to pre illness physical capabilities. Emphasis has recently been placed on finding innovative multi-disciplinary methods that can improve the care of elderly people who had suffered an acute illness. The aim of this prospective study is to assess the effect of mind-body therapy(including guided imagery, relaxation techniques, mediation and touch therapy) as as an adjunct to medical and physical rehabilitation in geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients,age 18 and above.
2. Getting standard rehabilitation therapy
3. Can fill an informed consent.

Exclusion Criteria:

1. Medically unstable patients (uncontrolled heart failure,rapid AF, severe infection, constant need of oxygen therapy).
2. Demented patients who are unable to fill an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
effect on quality of life | 1 year

SECONDARY OUTCOMES:
effect of treatment on rehabilitation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center; ,, Tel Aviv, Israel, Israel